CLINICAL TRIAL: NCT00137319
Title: An Evaluation of an Impedance Threshold Device (ITD) to Improve Hemodynamic Function During Orthostatic Challenge in Burn Patients
Brief Title: Impedance Threshold Device Tilt Study
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Aims of the study re-evaluated, did not justify allocation of resources.
Sponsor: United States Army Institute of Surgical Research (U.S. Federal Agency)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-04-016
Record Dates: First submitted 2005-08-25; First posted 2005-08-29 (Estimated); Last update posted 2015-07-22 (Estimated); Status verified 2015-07

CONDITIONS: Orthostatic Hypotension
Keywords: inspiratory impedance threshold device; blood pressure regulation; head-up tilt test; tilt table testing; burn injury; Burns
MeSH Terms: conditions — Hypotension, Orthostatic; Burns

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Impedance threshold device

SUMMARY:
This study will see if a special piece of equipment can help burn patients who have been in bed for a long time to get out of bed without feeling dizzy or faint.

DETAILED DESCRIPTION:
To measure stroke volume, cardiac output, arterial blood pressure and cerebral blood flow velocity in human patients while they undergo exposure to head-up tilt that is designed to test their tolerance to an orthostatic challenge.

ELIGIBILITY:
Inclusion Criteria:

* Military or civilian males or females between the ages of 18-65 years
* Burn injury with at least one unburned finger for Portapres measurement
* Minimum of 96 hours bedrest or physician directive to tilt

Exclusion Criteria:

* Age < 18 and > 65 years
* Facial burns when application of ITD device would cause further trauma
* Medical monitoring devices that preclude the use of the ITD
* Signs of cardiac abnormalities, autonomic dysfunction
* Chronic obstructive pulmonary disease (COPD), or any other respiratory limitations (ventilator dependent, intubated, tracheostomy) limiting use of ITD
* History of pre-syncopal/syncopal episodes or orthostatic hypotension
* History of atherosclerotic coronary heart disease
* Patients taking any kind of cardiovascular pressor medications
* Inability to obtain a Portapres pulse wave validated by blood pressure cuff with +/- 5mmHg diastolic blood pressure
* Unable to provide informed consent for self

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2004-10; Study Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
Inspiratory impedance during passive upright tilt will prevent orthostatic hypotension. | 1 hour

CONTACTS AND LOCATIONS:
Overall Officials: Travis Hedman, MPT, CPT, SP, Principal Investigator — US Army Institute of Surgical Research
Locations (1):
- US Army Institute of Surgical Research, Fort Sam Houston, Texas, United States

REFERENCES:
- [Background] Convertino VA, Idris A, Ratliff D, Ryan K, Doerr D, Lurie K. Use of an inspiratory impedance threshold valve increases cardiac output in human volunteers. Crit. Care Med. 30:A66, 2003